CLINICAL TRIAL: NCT01999205
Title: Moving To Business: Promoting Physical Activity and Reducing Sedentary Behavior in Office-based Companies in Finland (MTB)
Brief Title: Moving To Business: Promoting Physical Activity and Reducing Sedentary Behavior in Office-based Companies in Finland
Acronym: MTB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UKK Institute (Other)
Collaborators: Finnish Institute of Occupational Health (Other); Finnish Sports Confederation (Unknown); Päijät-Hämeen Liikunta ja urheilu ry (Unknown); Etelä-Karjalan Liikunta ja Urheilu ry (Unknown); Hämeen Liikunta ja Urheilu ry (Unknown)
Responsible Party: Principal Investigator, Minna Aittasalo, Docent, DSc, PT, Researcher, UKK Institute
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 175
Record Dates: First submitted 2013-11-01; First posted 2013-12-03 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Physical Activity; Sedentary Behavior; Work Ability
Keywords: workplace; intervention; physical activity; sedentary behavior; evaluation
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical activity promotion (Experimental): A nominated team in each participating company develops a plan to promote physical activity and to reduce sedentary behavior of the employees
  Interventions: Behavioral: Physical activity promotion

INTERVENTIONS:
Behavioral: Physical activity promotion — A nominated team in each participating company develops a plan to promote physical activity and to reduce sedentary behavior of the employees.

SUMMARY:
The participants are twelve small or middle-sized companies. Baseline information about the company's practices and employees' physical activity is collected in November 2013 with questionnaires and accelerometers. A team is nominated in each company to develop company's practices in relation to promoting physical activity and reducing sedentary behavior among employees. The teams are supported with materials and meetings and the opportunity to obtain physical activity services from the regional offices of the Finnish Sports Confederation. The development process is carried out in Fall 2013 and the actions to promote physical activity and to reduce sedentary behavior are implemented in the companies during spring and fall 2014. The follow-up evaluation with the same measures as at baseline will be conducted in November 2014 and depending on financing possibly also in November to assess the maintenance of the actions.

ELIGIBILITY:
Inclusion Criteria:

* companies: number of employees 15-150 (small or middle-sized)
* employees: all voluntary employees

Exclusion Criteria:

* companies: less than 15 or more than 150 employees
* employees: none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Physical activity and sedentary behavior | One year
  Change in the accelerometer-determined and self-reported (questionnaire) physical activity and sedentary behavior of the employees from baseline to 12 months.

SECONDARY OUTCOMES:
Work ability | One year
  Change in the self-reported work ability (questionnaire scale from 0 to 10) from baseline to 12 months.

OTHER OUTCOMES:
Employees' participation in staff physical activity | One year
  Change in employees' self-reported (questionnaire) participation in staff physical activity from baseline to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Minna Aittasalo, DSc, Principal Investigator — UKK Institute
Locations (1):
- The UKK Institute for Health Promotion Research, Tampere, Pirkanmaa, Finland

REFERENCES:
- [Derived] Aittasalo M, Livson M, Lusa S, Romo A, Vaha-Ypya H, Tokola K, Sievanen H, Manttari A, Vasankari T. Moving to business - changes in physical activity and sedentary behavior after multilevel intervention in small and medium-size workplaces. BMC Public Health. 2017 Apr 17;17(1):319. doi: 10.1186/s12889-017-4229-4. PMID 28415993
- See also: Related Info — http://www.ukkinstituutti.fi